CLINICAL TRIAL: NCT07158333
Title: Mobile Cardiac Telemetry (MCT) Study
Status: Completed | Type: Observational
Sponsor: Baxter Healthcare Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: BXU607689
Record Dates: First submitted 2025-08-28; First posted 2025-09-05 (Actual); Last update posted 2025-11-12 (Actual); Status verified 2025-11

CONDITIONS: Healthy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (1):
- MCT device subjects: All subjects are provided MCT system
  Interventions: Device: Mobile Cardiac Telemetry (MCT System)

INTERVENTIONS:
Device: Mobile Cardiac Telemetry (MCT System) — MCT System without data transmission

SUMMARY:
This study will be a single center, single arm, open-label, prospective study to evaluate adhesive performance of the Bardy Diagnostics' (BardyDx) MCT Patch up to 30 days of wear.

ELIGIBILITY:
Inclusion Criteria:

Each subject must meet the following criteria to be enrolled in this study:

1. Subject is ≥18 years of age.
2. Completes the consent process as required.
3. Subject can speak and read English fluently.
4. Subject is willing to allow shaving of device application area, as required.
5. Subject is willing and able to take photos of the application area before, during, and immediately after wear of each Adhesive Patch

Exclusion Criteria:

1. Unable to comply with the study protocol and instructions for wearing the MCT Patch for up to 30 days.
2. Geographically located such that they cannot have the initial MCT Patch placed by PI or designee.
3. Any breached or compromised skin, skin rash, irritation or infection over the sternum (prior to the initial application) as reported by the subject and/or observed by the PI during initial application.
4. Had any sternal incision or wound within 3 months prior to the date of enrolment.
5. Subjects with sensitive skin or known skin conditions, including known allergies.
6. Subjects with scheduled cardioversion during the data collection period.
7. Subjects with a scheduled electronic imaging (including magnetic resonance imaging) during the data collection period.
8. Subject has known cardiac arrhythmia conditions (Note: The PI will assess the subject during initial screening. If an arrhythmia is discovered during the subject will be deemed ineligible for participation in the study).

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: A total of 10 healthy evaluable subjects (wearing and returning the test article) consisting of at least 5 males and 5 females is the desired sample size.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2025-08-05 (Actual); Primary Completion 2025-09-12 (Actual); Study Completion 2025-09-12 (Actual)

PRIMARY OUTCOMES:
Cumulative wear time | 30 days
  as measured by ECG readability sufficient for identification of the P and QRS waves; the total readable duration summed from each patch, measured from the start of the first day to the end

SECONDARY OUTCOMES:
Subject Self-Reported Log & Subject Survey of the MCT Patch after 30 days | 30 days
  skin and adhesive comfort, and device stability and skin contact
Adverse events of relevance, including potential skin damage due to repeated removal and reapplication of the MCT Patch as determined by Investigator/designee from subject assessments including Subject Logs, Subject Surveys and photos. | From enrollment to end of study at 30 days.

CONTACTS AND LOCATIONS:
Locations (1):
- Orange County Research Center, Lake Forest, California, United States